CLINICAL TRIAL: NCT02521194
Title: Is Inpatient Occupational Therapy Perceived to be Beneficial by the Palliative Patient and Caregiver?
Brief Title: Occupational Therapy in Palliative Care
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI requested
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-0350
Record Dates: First submitted 2015-08-10; First posted 2015-08-13 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Advanced Cancers
Keywords: Advanced Cancers; Inpatient occupational therapy; Questionnaire; Survey
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caregiver Questionnaire (Experimental): Questionnaire completion regarding opinion on the inpatient occupational therapy session person being cared for received.
  Interventions: Behavioral: Questionnaire
- Patient Questionnaire (Experimental): Questionnaire completion regarding opinion of the inpatient occupational therapy session patient received.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire completion regarding opinion of the inpatient occupational therapy session patient received.
  Other Names: Survey

SUMMARY:
The goal of this research study is to learn if inpatient occupational therapy can help patients in the Palliative Care Unit (PCU).

DETAILED DESCRIPTION:
Caregivers Consent:

If you agree to take part in this study, you will complete a questionnaire about your opinion on the inpatient occupational therapy session the patient (person you are caring for) received. It should take about 10 minutes to complete the questionnaire. You will be left alone in a room to complete the questionnaire.

Length of Study:

Your participation on this study will be over after you complete the questionnaire.

This is an investigational study.

50 patients and up to 50 caregivers will take part in this study. All will be enrolled at MD Anderson.

Patients Consent:

If you agree to take part in this study, you will complete a questionnaire about your opinion of the inpatient occupational therapy session you just had. The questionnaire should take about 10 minutes to complete. You will be left alone in the room to complete the questionnaire.

Length of Study:

You participation on this study will be over after you complete the questionnaire.

This is an investigational study.

50 patients and up to 50 caregivers will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have an inpatient occupational therapy (OT) order and be able to tolerate an OT session as judged by the attending physician
2. Patients with cancer admitted to inpatient acute palliative care unit
3. Caregiver participation is optional, but must be identified as the primary caregiver in order to complete the Caregiver Satisfaction Survey.
4. Caregiver (if participating) must be present during the session.
5. Patient (and caregiver (if participating) must be 18 years of age or older.
6. Both patient (and caregiver if participating) must be able to understand, read, write and speak English.
7. Both patient and caregiver (if participating) must sign an Informed Consent Form.

Exclusion Criteria:

1. Patients or caregivers with physical limitations (visual or motor impairment) causing inability to read, complete or sign the consent form and survey.
2. Patients or caregivers who the attending physician deems unable to participate due to poor cognitive capacity or acute physical distress.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2015-11-13 (Actual); Primary Completion 2020-01-05 (Actual); Study Completion 2020-01-05 (Actual)

PRIMARY OUTCOMES:
Satisfaction Rate of Inpatient Occupational Therapy Session | 1 day
  Satisfaction rate defined as the percentage of patients that "strongly agree" or "agree" after inpatient occupational session as being beneficial.

CONTACTS AND LOCATIONS:
Overall Officials: Paul W. Walker, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org